CLINICAL TRIAL: NCT01133379
Title: Evaluation of the Efficacy of Two Potassium Oxalate Containing Mouthrinses for Relieving Dentinal Hypersensitivity
Brief Title: Tooth Sensitivity Relief by Two Mouthrinses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KOXDHY0001
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PO-019 (Experimental): 1.40% Potassium Oxalate Sensitive Mouthwash without fluoride (12027-019)
  Interventions: Device: 12027-019
- PO-020 (Experimental): 1.40% Potassium Oxalate Sensitive Mouthwash with fluoride (12027-020)
  Interventions: Device: 12027-020
- PO-021 (Sham Comparator): Vehicle Control Mouthrinse (without potassium oxalate and without fluoride) (12027-021)
  Interventions: Device: 12027-021

INTERVENTIONS:
Device: 12027-019 — Rinse with 10 mL for 60 seconds twice daily after brushing in your usual manner for 1 minute using at least a one-inch strip of the assigned toothpaste.
  Other Names: 1.40% Potassium Oxalate Sensitive Mouthwash without fluoride
  Arms: PO-019
Device: 12027-020 — Rinse with 20 mL for 60 seconds twice daily after brushing in your usual manner for 1 minute using at least a one-inch strip of the assigned toothpaste.
  Other Names: 1.40% Potassium Oxalate Sensitive Mouthwash with fluoride
  Arms: PO-020
Device: 12027-021 — Rinse with 10 mL for 60 seconds twice daily after brushing in your usual manner for 1 minute using at least a one-inch strip of the assigned toothpaste
  Other Names: Vehicle Control Mouthrinse
  Arms: PO-021

SUMMARY:
This study is for people with sensitive teeth and involves going to the dentist for 6 visits over 8 weeks. During the first 2 weeks, everyone will just brush their teeth two times a day with the fluoride toothpaste provided.

Then you will be assigned to a mouthwash group if you qualify to continue in the study. Two groups will get mouthwash with a certain amount of an experimental ingredient and one group will get a mouthwash with no experimental ingredients. You will have an equal chance of being assigned to any one of the three groups.

For the next 6 weeks, you will rinse with your assigned mouthwash after brushing. A dentist will look at your mouth, teeth, tongue and gums and check for sensitive teeth. The investigators will see if the mouthwash helps to reduce tooth sensitivity during the study.

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel group, single center, controlled clinical trial design. Approximately 200 generally healthy adults meeting the necessary inclusion/exclusion criteria will be enrolled so that 180 subjects (60 per treatment group) would reasonably be expected to complete the study. Subjects will have their oral soft/hard tissues assessed and will be evaluated for sensitivity levels at Screening (visit 1), Baseline (visit 2), Week 1, Week 2, Week 4 & Week 6. During the first two weeks of the study, subjects will be instructed to brush their teeth for one minute in their usual manner, twice daily using the provided standard fluoride toothpaste. Subjects will return for the Baseline exam and, upon qualification with entry criteria, will be assigned to one of three treatment groups. Qualified subjects will be instructed to brush their teeth two times daily for one minute in their usual manner using the provided standard fluoride toothpaste. Subjects will be instructed to rinse twice daily, after brushing, with the provided mouthrinse for 60 seconds using 10 ml or 20 ml (depending on the treatment group), for 6 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age in good general and oral health without any known allergy to commercial dental products or cosmetics.
* Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial
* Willingness to use the assigned products according to instructions, availability for appointments, and likelihood of completing the clinical trial.
* A minimum of 2 natural premolars, canines, and/or incisors teeth with decay-free scorable facial/buccal surfaces which must present cervical abrasion, and/or erosion and/or gingival recession.
* A minimum of two eligible teeth (premolars, canines and/or incisors) with a Screening (-2 weeks Baseline) and Baseline tactile sensitivity score between 10 - 50 grams after application of the Yeaple probe and a cold air stimulus VAS score of 30 - 80 mm on a 100 mm VAS scale will be followed as study teeth during the trial.
* No more than two eligible teeth per quadrant each separated by 2 other teeth must be selected.Absence of significant oral soft tissue pathology, based on the dentist's visual examination and at the discretion of the investigator.
* Adequate oral hygiene (i.e. brush teeth daily and exhibit no signs of oral neglect).
* Absence of severe marginal gingivitis, moderate/advanced periodontitis (ADA Type III, IV) based on a clinical examination and discretion of the Investigator.
* Absence of extensive supragingival calculus.

Exclusion Criteria:

* Volunteers who report history or presence of kidney disorders, kidney stones, eating disorders, uncontrolled GERD, excessive dietary or environmental exposure to acids, or other systemic conditions that are predisposing to dentinal hypersensitivity.
* Volunteers with chronic medical debilitating disease associated with constant or intermittent episodes of daily pain.
* Long-term daily use (≥ 7 consecutive days) of analgesics and any other drugs that at the discretion of the Investigator would compromise the response of the hypersensitivity assessments.
* Volunteers who have been using any home-care bleaching, whitening products or have had a professional bleaching treatment within 4 weeks of the Screening visit.
* Use of desensitizing agents whether prescribed or over-the-counter within eight weeks prior to screening visit (any sensitivity toothpastes such as Crest Sensitivity, Sensodyne, Crest Pro-Health, Colgate Sensitivity Relief, any mouthwash and oral care products used for the treatment of dentinal hypersensitivity).
* Volunteers who during the study will receive dental treatment which may affect their dentinal hypersensitivity condition (i.e. oral prophylaxis). Emergency treatment will be allowed.
* Those requiring antibiotic premedication prior to invasive dental procedures.
* Participation in a dental clinical trial involving oral care products within the past 30 days.
* Women who are pregnant, nursing or plan to become pregnant during the course of the study.
* Teeth that are grossly carious, orthodontically banded, abutment teeth for fixed or removable prostheses, crowned teeth, or third molars will not be included in the study.
* Periodontal surgery and orthodontic treatment within previous 3 months.
* Extensive restorative treatment (i.e. extensively restored teeth or teeth with restoration(s) extending into the test area) at the discretion of the Investigator.
* Dental prophylaxis within 2 weeks prior to Screening visit.
* Teeth or periodontium with pathology or defect likely to cause pain.
* Teeth with clinical mobility > grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hee, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- BioSci Research America, Inc., Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 12027-021 (Vehicle Control): Vehicle Control Mouth Rinse (without Potassium Oxalate and without Fluoride) (10 mL)
- 12027-019: 1.40% Potassium Oxalate Sensitive Mouth Rinse without Fluoride (10 mL)
- 12027-020: 1.40% Potassium Oxalate Sensitive Mouth Rinse with Fluoride (20 mL)
Period: Overall Study
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Started | 58 | 58 | 58
Completed | 57 | 56 | 56
Not Completed | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020 | Total
Number analyzed (Participants) | 58 | 58 | 58 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (11.36) | 33.9 (10.98) | 35.8 (11.98) | 35.0 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 42 | 127
  Male | 15 | 16 | 16 | 47
Region of Enrollment [Number; unit: participants]
  USA | 58 | 58 | 58 | 174

OUTCOME MEASURES:

1. Primary Outcome: Mean Tactile Sensitivity Score at Week 6
Description: Tooth sensitivity was measured using a Yeaple probe. The force at which discomfort was felt by the participant was recorded on a scale of 10-80 grams. The score for each participant was calculated by averaging the scores for all study teeth for that participant, at each visit.
Time Frame: 6 Weeks
Population: Analysis was based on the Intent-to-Treat Analysis Set, which included all randomized participants who used at least one dose of the study product and had baseline and at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 57 | 56 | 56
grams | 37.91 (3.342) | 36.77 (3.362) | 30.16 (3.362)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; The null hypothesis was no difference in mean outcome between treatment groups. The alternative hypothesis was a difference in mean outcome between treatment groups; Test type: Superiority or Other; p = 0.811, ANCOVA — Per statistical analysis plan, if experimental rinse (12027-019) was better than vehicle control at Week 6 (p<0.05), testing for 12027-019 versus vehicle control proceeded to Week 4. Family-wise error rate was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-10.5 to 8.24], Standard Error of Mean 4.750
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.105, ANCOVA — Per statistical analysis plan, if experimental rinse (12027-020) was better than vehicle control at Week 6 (p<0.05), testing for 12027-020 versus vehicle control proceeded to Week 4. Family-wise error rate was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = -7.75, 95% CI 2-sided [-17.1 to 1.63], Standard Error of Mean 4.750

2. Primary Outcome: Mean Tactile Sensitivity Score at Week 4
Description: as for outcome 1
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 57 | 56 | 56
grams | 30.58 (2.793) | 31.69 (2.809) | 25.66 (2.809)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.779, ANCOVA — Per statistical analysis plan, if experimental rinse (12027-019) was better than vehicle control at Week 4 (p<0.05), testing for 12027-019 versus vehicle control proceeded to Week 2. Family-wise error rate was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [-6.72 to 8.95], Standard Error of Mean 3.969
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.217, ANCOVA — Per statistical analysis plan, if experimental rinse (12027-020) was better than vehicle control at Week 4 (p<0.05), testing for 12027-020 versus vehicle control proceeded to Week 2. Family-wise error rate was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = -4.92, 95% CI 2-sided [-12.8 to 2.92], Standard Error of Mean 3.969

3. Primary Outcome: Mean Tactile Sensitivity Score at Week 2
Description: as for outcome 1
Time Frame: 2 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 58 | 57 | 57
grams | 22.27 (1.838) | 22.59 (1.849) | 18.28 (1.849)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.904, ANCOVA — Per statistical analysis plan, if experimental rinse (12027-019) was better than vehicle control at Week 2 (p<0.05), testing for 12027-019 versus vehicle control proceeded to Week 1. Family-wise error rate was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-4.84 to 5.47], Standard Error of Mean 2.613
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.129, ANCOVA — Per statistical analysis plan, if experimental rinse (12027-020) was better than vehicle control at Week 2 (p<0.05), testing for 12027-020 versus vehicle control proceeded to Week 1. Family-wise error rate was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = -3.99, 95% CI 2-sided [-9.15 to 1.17], Standard Error of Mean 2.613

4. Primary Outcome: Mean Tactile Sensitivity Score at Week 1
Description: as for outcome 1
Time Frame: 1 Week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 58 | 58 | 58
grams | 15.99 (0.944) | 15.04 (0.941) | 15.03 (0.941)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.477, ANCOVA — The significance threshold was 0.05. Family-wise error rate was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-3.59 to 1.69], Standard Error of Mean 1.336
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.472, ANCOVA — The significance threshold was 0.05. Family-wise error rate was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-3.60 to 1.67], Standard Error of Mean 1.336

5. Secondary Outcome: Mean Tactile Sensitivity VAS Score at Week 1
Description: Tooth sensitivity was measured using a Visual Analogue Scale (VAS). At each visit, participants rated their perception of the pain/discomfort experienced from the Yeaple probe by marking a single vertical line on a VAS scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm. The investigator recorded a VAS score of 0 mm for participants who did not experience discomfort at the maximum force of 80 grams. The score for each participant was calculated by averaging the scores for all study teeth for that participant.
Time Frame: 1 Week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 58 | 58 | 58
units on a scale (mm) | 40.09 (1.926) | 39.61 (1.927) | 39.27 (1.926)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.860, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-5.86 to 4.90], Standard Error of Mean 2.726
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.763, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-6.20 to 4.55], Standard Error of Mean 2.723

6. Secondary Outcome: Mean Tactile Sensitivity VAS Score at Week 2
Description: as for outcome 5
Time Frame: 2 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 58 | 57 | 57
units on a scale (mm) | 37.69 (2.010) | 35.71 (2.028) | 34.79 (2.027)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.488, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-7.62 to 3.66], Standard Error of Mean 2.856
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.311, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -2.90, 95% CI 2-sided [-8.54 to 2.73], Standard Error of Mean 2.854

7. Secondary Outcome: Mean Tactile Sensitivity VAS Score at Week 4
Description: as for outcome 5
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 57 | 56 | 56
units on a scale (mm) | 31.06 (2.448) | 29.25 (2.469) | 32.97 (2.469)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.604, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-8.68 to 5.06], Standard Error of Mean 3.478
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.583, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = 1.91, 95% CI 2-sided [-4.95 to 8.78], Standard Error of Mean 3.477

8. Secondary Outcome: Mean Tactile Sensitivity VAS Score at Week 6
Description: as for outcome 5
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 57 | 56 | 56
units on a scale (mm) | 25.50 (2.541) | 24.80 (2.563) | 26.86 (2.563)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.847, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-7.83 to 6.43], Standard Error of Mean 3.610
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.708, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = 1.36, 95% CI 2-sided [-5.77 to 8.48], Standard Error of Mean 3.610

9. Secondary Outcome: Mean Cold Air Stimulus VAS Score at Week 1
Description: Tooth sensitivity was measured using a Cold Air Stimulus. When being assessed, participants rated their perception of the pain/discomfort experienced when cold air was directed at the exposed root of each tooth by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm. The score for each participant was calculated by averaging the scores for all study teeth for that participant.
Time Frame: 1 Week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 58 | 58 | 58
units on a scale (mm) | 44.18 (1.894) | 41.72 (1.893) | 40.30 (1.893)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.360, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air VAS score; Mean Difference (Final Values) = -2.46, 95% CI 2-sided [-7.75 to 2.83], Standard Error of Mean 2.678
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.149, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air VAS score; Mean Difference (Final Values) = -3.88, 95% CI 2-sided [-9.17 to 1.41], Standard Error of Mean 2.679

10. Secondary Outcome: Mean Cold Air Stimulus VAS Score at Week 2
Description: as for outcome 9
Time Frame: 2 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 58 | 57 | 57
units on a scale (mm) | 40.56 (2.277) | 37.95 (2.296) | 36.90 (2.296)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.421, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air VAS score; Mean Difference (Final Values) = -2.61, 95% CI 2-sided [-9.00 to 3.78], Standard Error of Mean 3.235
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.260, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air VAS score; Mean Difference (Final Values) = -3.66, 95% CI 2-sided [-10.0 to 2.73], Standard Error of Mean 3.235

11. Secondary Outcome: Mean Cold Air Stimulus VAS Score at Week 4
Description: as for outcome 9
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 57 | 56 | 56
units on a scale (mm) | 31.92 (2.534) | 31.87 (2.556) | 30.63 (2.555)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.989, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air VAS score; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-7.16 to 7.06], Standard Error of Mean 3.601
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.721, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air VAS score; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-8.39 to 5.82], Standard Error of Mean 3.599

12. Secondary Outcome: Mean Cold Air Stimulus VAS Score at Week 6
Description: as for outcome 9
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 57 | 56 | 56
units on a scale (mm) | 26.61 (2.597) | 25.40 (2.619) | 26.28 (2.618)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.743, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air VAS score; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-8.50 to 6.07], Standard Error of Mean 3.690
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.928, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air VAS score; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-7.61 to 6.95], Standard Error of Mean 3.688

13. Secondary Outcome: Global Subjective VAS Score at Week 1
Description: At Week 1, participants rated their perception of the pain/discomfort experienced by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. Participants were instructed as follows: "Please rate the intensity of the pain/discomfort you have experienced in the last week when drinking cold/hot beverages and/or foods, eating sweet and sour foods, breathing cold air, brushing your teeth or performing any habits/behaviors that solicit your dentinal hypersensitivity pain/discomfort since you first started using the product." The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm.
Time Frame: 1 Week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 58 | 58 | 58
units on a scale (mm) | 47.54 (1.675) | 48.51 (1.676) | 47.28 (1.677)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.683, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline global subjective VAS score; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [-3.71 to 5.65], Standard Error of Mean 2.369
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.914, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline global subjective VAS score; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-4.94 to 4.42], Standard Error of Mean 2.371

14. Secondary Outcome: Global Subjective VAS Score at Week 2
Description: At Week 2, participants rated their perception of the pain/discomfort experienced by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. Participants were instructed as follows: "Please rate the intensity of the pain/discomfort you have experienced in the last two weeks when drinking cold/hot beverages and/or foods, eating sweet and sour foods, breathing cold air, brushing your teeth or performing any habits/behaviors that solicit your dentinal hypersensitivity pain/discomfort since you first started using the product." The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm.
Time Frame: 2 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 58 | 57 | 57
units on a scale (mm) | 44.12 (2.108) | 37.93 (2.128) | 38.02 (2.129)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.040, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline global subjective VAS score; Mean Difference (Final Values) = -6.19, 95% CI 2-sided [-12.1 to -0.27], Standard Error of Mean 2.994
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.043, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline global subjective VAS score; Mean Difference (Final Values) = -6.10, 95% CI 2-sided [-12.0 to -0.18], Standard Error of Mean 2.997

15. Secondary Outcome: Global Subjective VAS Score at Week 4
Description: At Week 4, participants rated their perception of the pain/discomfort experienced by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. Participants were instructed as follows: "Please rate the intensity of the pain/discomfort you have experienced in the last two weeks when drinking cold/hot beverages and/or foods, eating sweet and sour foods, breathing cold air, brushing your teeth or performing any habits/behaviors that solicit your dentinal hypersensitivity pain/discomfort since you first started using the product." The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 57 | 56 | 56
units on a scale (mm) | 35.92 (2.480) | 33.60 (2.503) | 31.85 (2.504)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.511, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline global subjective VAS score; Mean Difference (Final Values) = -2.32, 95% CI 2-sided [-9.27 to 4.64], Standard Error of Mean 3.522
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.250, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline global subjective VAS score; Mean Difference (Final Values) = -4.07, 95% CI 2-sided [-11.0 to 2.89], Standard Error of Mean 3.526

16. Secondary Outcome: Global Subjective VAS Score at Week 6
Description: At Week 6, participants rated their perception of the pain/discomfort experienced by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. Participants were instructed as follows: "Please rate the intensity of the pain/discomfort you have experienced in the last two weeks when drinking cold/hot beverages and/or foods, eating sweet and sour foods, breathing cold air, brushing your teeth or performing any habits/behaviors that solicit your dentinal hypersensitivity pain/discomfort since you first started using the product." The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Number analyzed (Participants) | 57 | 56 | 56
units on a scale (mm) | 31.15 (2.593) | 26.74 (2.617) | 25.31 (2.619)
Statistical Analysis 1: Comparison: 12027-021 (Vehicle Control) vs 12027-019; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.233, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline global subjective VAS score; Mean Difference (Final Values) = -4.41, 95% CI 2-sided [-11.7 to 2.86], Standard Error of Mean 3.684
Statistical Analysis 2: Comparison: 12027-021 (Vehicle Control) vs 12027-020; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.115, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline global subjective VAS score; Mean Difference (Final Values) = -5.84, 95% CI 2-sided [-13.1 to 1.44], Standard Error of Mean 3.687

ADVERSE EVENTS:
Time Frame: Day 43 ± 3 days, + 30 days for serious adverse events.
Description: Adverse events were systematically collected at each study visit through Visit 6 (Day 43 ± 3 days). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | 12027-021 (Vehicle Control) | 12027-019 | 12027-020
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator agreed not to publish the study results without prior sponsor approval.